CLINICAL TRIAL: NCT01473082
Title: Comparison of Proximal Femoral Nail Antirotation (PFNA) Versus PFNA Augmentation for the Treatment of Closed Unstable Trochanteric Fractures - A Randomized-controlled Trial
Brief Title: Proximal Femoral Nail Antirotation (PFNA) Versus PFNA Augmentation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PFNA augmented
Record Dates: First submitted 2011-11-10; First posted 2011-11-17 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2018-07

CONDITIONS: Hip Fractures; Closed Fracture of Hip
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PFNA (Active Comparator): Proximal Femoral Nail Antirotation (PFNA Synthes)
  Interventions: Device: PFNA (Synthes)
- PFNA Augmentation (Active Comparator): Proximal Femoral Nail Antirotation PFNA Augmentation (Synthes) with Traumacem V+ Synthes
  Interventions: Device: PFNA Augmentation (Synthes)

INTERVENTIONS:
Device: PFNA Augmentation (Synthes) — Proximal Femoral Nail Antirotation (PFNA) Augmentation (with Traumacem V+)
  Other Names: PFNA Augmentation (Synthes) length 240 mm; PFNA Augmentation (Synthes) small length 200 mm; PFNA Augmentation (Synthes) xs length 170 mm; PFNA Augmentation (Synthes) long lengths 300-420 mm
  Arms: PFNA Augmentation
Device: PFNA (Synthes) — Proximal Femoral Nail Antirotation (PFNA)
  Other Names: PFNA length 240 mm; PFNA small length 200 mm; PFNA xs length 170 mm; PFNA long lengths 300-420 mm
  Arms: PFNA

SUMMARY:
The purpose of this study is to evaluate whether patients with trochanteric fractures being treated with a Proximal Femoral Nail Antirotation (PFNA) and augmentation can better be mobilized than patients without augmentation.

DETAILED DESCRIPTION:
To avoid the pain-causing relative movement between implant and bone, surgical techniques and devices allowing augmentation of the femoral head have recently been developed. Biomechanical studies showed that augmentation leads to a better axial stability and pull-out strength. In clinical practice, this might facilitate early mobilization and full weight-bearing with less pain. The purpose of this study is therefore to evaluate whether patients with trochanteric fractures being treated with a PFNA and augmentation can better be mobilized than patients without augmentation. In particular, it will be measured whether patients with a PFNA Augmentation can walk faster than the non-augmented patients, measured with the Timed up and Go test.

ELIGIBILITY:
Inclusion Criteria:

* Age 75 years and older
* Closed unstable trochanteric fracture: AO 31 - A2 and A3
* Low energy trauma (e.g.fall from standing height)
* Definitive fracture fixation within 72 hrs. after admission
* Indication for PFNA fixation (with or without augmentation)
* Ability to walk independently (walking aids are allowed) prior to injury
* Signed written informed consent and agreement to attend the planned FUs
* Able to understand and read country national language at an elementary level

Exclusion Criteria:

* Pathologic fracture
* Polytrauma
* Any additional fracture
* Open fracture
* Recent history of substance abuse (ie, recreational drugs, alcohol) that would preclude reliable assessment
* Active malignancy defined as history of invasive malignancy, except if the patient has received treatment and displayed no clinical signs and symptoms for at least five years
* ASA class V and VI
* Any implant at the same hip
* Hemiplegia
* Patients with legal guardian
* Patients who have participated in any other device or drug related clinical trial that could influence the results of the present study within the previous month
* Fractures and injuries opening into the articulation and vascular structure
* Infection
* Patients with clotting disorders
* Patients with severe cardiac and / or pulmonary insufficiency
* Patients with known hypersensitivity or allergy to any of the components of Traumacem V+ cement (Polymethyl methacrylate / acrylate, zirconium dioxide, hydroxyapatite,benzoyl peroxide, methyl methacrylate,hydroquinone, N,N-dimethyl-p-toluidine)
* Perforation of the femoral head into the joint with the guide wire used for the PFNA blade
* Risk of potential leakage into the joint identified by using contrast fluid (PFNA Augmentation group only)
* Intraoperative decision to use implants other than PFNA

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 251 (Actual)
Dates: Start 2012-02; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Mobility measured with the "timed up & go"-test during hospital stay. | 5 to 7 days postoperative
  The TUG measures the time (in seconds) that it takes for an individual to rise from an armchair (chair seat height = 45 cm / 1.5 feet), walk 3 meters (= 10 feet) to a line drawn on the floor, turn around and return to the chair. The time is measured from a seated position (back against the backrest) with a stopwatch started on the command "ready - go" and stopped when the seat position is reached again. Patient-perceived pain and exertion will be assessed after the test.

SECONDARY OUTCOMES:
Description of surgical details as surgery time and fluoroscopy time, and of augmentation details (PFNA Augmentation group only). | Intraoperative
Pain | one year
  Pain, measured with the Numerical Rating Scale (NRS) and use of pain medication postoperative.
Duration of hospital stay | one year
Walking ability | one year
  Parker Mobility Score
Return to pre-fracture residential status | one year
Timed up & go-test at follow-ups | one year
  The TUG measures the time (in seconds) that it takes for an individual to rise from an armchair (chair seat height = 45 cm / 1.5 feet), walk 3 meters (= 10 feet) to a line drawn on the floor, turn around and return to the chair. The time is measured from a seated position (back against the backrest) with a stopwatch started on the command "ready - go" and stopped when the seat position is reached again.
Quality of life | one year
  EuroQol-5D
Local adverse events and revision rate | one year
  Implant / surgery, bone / fracture, soft tissue of the musculoskeletal system, wound related adverse events
Systemic adverse events | one year
Implant migration | one year
  Measured at the CT in a subgroup only
Mortality | one year
Fracture risk prior to injury | 1 week prior to operation
  Measured with the Fracture Risk Assessment Tool (FRAX)
Functional independence | 1 week prior to operation
  Measured with the Barthel Index
Comorbidity | 1 week prior to operation
  Charlson Comorbidiy Index

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Faeh, Study Director — AO Clinical Investigation and Documentation, Davos, Switzerland; Christian Kammerlander, MD, Principal Investigator — Medical University of Innsbruck, Austria
Locations (9):
- Medical University of Innsbruck, Innsbruck, Austria
- KUL Univ. Ziekenhuizen Leuven, Leuven, Belgium
- Germany (3):
  - BGU Tübingen, Tübingen
  - University of Ulm, Ulm
  - Sophien und Hufeland Klinikum GmbH, Weimar
- Hadassah Medical Organization, Jerusalem, Israel
- Sykehuset i Vestfold HF Tønsberg, Tønsberg, Norway
- Switzerland (2):
  - Cantonal Hospital Lucerne, Lucerne
  - City Hospital Waid, Zurich

REFERENCES:
- [Result] Kammerlander C, Hem ES, Klopfer T, Gebhard F, Sermon A, Dietrich M, Bach O, Weil Y, Babst R, Blauth M. Cement augmentation of the Proximal Femoral Nail Antirotation (PFNA) - A multicentre randomized controlled trial. Injury. 2018 Aug;49(8):1436-1444. doi: 10.1016/j.injury.2018.04.022. Epub 2018 Apr 22. PMID 29724590